CLINICAL TRIAL: NCT01037985
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, WITHIN-SUBJECT CONTROLLED STUDY TO EVALUATE EFFICACY AND SAFETY OF EXC 001 FOR THE AMELIORATION OF SCARRING OF THE SURGICAL INCISION IN SUBJECTS UNDERGOING AN ELECTIVE ABDOMINOPLASTY
Brief Title: Safety and Efficacy Study of EXC 001 to Improve the Appearance of Scars in Subjects Undergoing Elective Abdominoplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: EXC 001-202; B5301010 (Other: Alias Study Number)
Record Dates: First submitted 2009-12-21; First posted 2009-12-23 (Estimated); Results first posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-06

CONDITIONS: Scar Prevention
Keywords: Scarring; Cicatrix; Fibrosis; Pathologic Process
MeSH Terms: conditions — Cicatrix; Fibrosis; Pathologic Processes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EXC 001 (Experimental)
  Interventions: Drug: EXC 001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EXC 001 — Multiple intradermal injections of EXC 001 and placebo
  Arms: EXC 001
Drug: Placebo — Multiple intradermal injections of EXC 001 and placebo
  Arms: Placebo

SUMMARY:
This study will compare how well EXC 001 works versus placebo in reducing the appearance of scars in subjects undergoing elective abdominoplasty. The study will also evaluate the safety of EXC 001 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have sufficient excess abdominal tissue to qualify for a standard elective abdominoplasty
* Subject has chosen to have an elective abdominoplasty
* Medically healthy with normal screening results
* Subjects must not be pregnant or lactating

Exclusion Criteria:

* Females who are currently pregnant or pregnant during the 12 months prior to inclusion in the study, or lactating
* Participation in another clinical trial within 30 days prior to the start of the study
* Any other condition or prior therapy, which, in the opinion of the PI, would make the subject unsuitable for this study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12-03 (Actual); Primary Completion 2010-07-07 (Actual); Study Completion 2010-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Scripps medical, La Jolla, California
  - Northwestern University,Division of Plastic Surgery, Chicago, Illinois
  - Barnes Jewish West County Hospital, St Louis, Missouri
  - Body Aesthetic Plastic Surgery, St Louis, Missouri
  - Jewell Plastic Surgery Center, Eugene, Oregon
  - Connall Consmetic Surgery, Tualatin, Oregon

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EXC001-202&StudyName=Safety%20and%20Efficacy%20Study%20of%20EXC%20001%20to%20Improve%20the%20Appearance%20of%20Scars%20in%20Subjects%20Undergoing%20Elective%20Abdominoplasty%0A

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who had chosen and qualified (sufficient excess abdominal tissue) for a standard elective abdominoplasty were recruited in this study. Study had 2 parts- Part A and B. Participants with negative skin sensitization in Part A (skin testing) were assigned to Part B (abdominoplasty surgery) of the study.
Groups:
- EXC 001 (PF-0647387) During Part A: In Part A participants received 2 intradermal injections on lower back of EXC 001 at a dose of 5 milligram (mg) on Day 1 and 21. Third 5 mg intradermal injection of EXC 001 was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery. The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until day of surgery in Part B.
- EXC 001 (PF-0647387) + Placebo During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent abdominoplasty surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear centimeter (cm) to a 6 cm section of both sides of abdominoplasty incision on one side of the midline and 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of abdominoplasty incision on another side of the midline, at Week 2, 5, 8, and 11 after the surgical incision was closed.
Period: Part A: Skin Testing (50 Days)
Arm/Group | EXC 001 (PF-0647387) During Part A | EXC 001 (PF-0647387) + Placebo During Part B
Started | 41 | 0
Completed | 37 | 0
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Physician Decision | 1 | 0
Period: Part B:Abdominoplasty Surgery (24 Weeks)
Arm/Group | EXC 001 (PF-0647387) During Part A | EXC 001 (PF-0647387) + Placebo During Part B
Started | 0 (Participants who tested negative for skin sensitization proceeded to Part B of the study. .) | 37 (Participants who completed Part A of the study and were negative for skin sensitization.)
Treated | 0 | 33
Completed | 0 | 32
Not Completed | 0 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Positive Skin Sensitization | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Groups:
- All Enrolled Participants: All participants who were enrolled in the study.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (4.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Expert Panel Scar Assessment Score at Week 12: Part B
Description: Scar assessment by an expert panel was done on blinded photographs using 100 millimeter (mm) visual analog scale (VAS) where a score of 0 = best possible scar and a score of 100 = worst possible scar. A pair of photographs for each participant were presented and evaluated 3 times by an expert panel.
Time Frame: Week 12
Population: Completer population included all participants who had missed not more than 1 dose of study drug, had the Week 12 assessment and non-missing data for VAS scar assessment score.
Measure: Mean (Standard Deviation); unit: millimeter
Groups:
- EXC 001 (PF-0647387) During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent abdominoplasty surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of abdominoplasty incision on one side of the midline at Week 2, 5, 8, and 11 after the surgical incision was closed.
- Placebo During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent abdominoplasty surgery on Day 1 and then received 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of abdominoplasty incision on another side of the midline, at Week 2, 5, 8, and 11 after the surgical incision was closed.
Arm/Group | EXC 001 (PF-0647387) During Part B | Placebo During Part B
Number analyzed (Participants) | 32 | 32
millimeter | 37.8 (12.96) | 42.1 (12.52)
Statistical Analysis 1: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Within participant treatment difference was assessed between the treatment regimens each participant received (EXC 001 minus placebo); Test type: Superiority; p = 0.168, t-test, 2 sided; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-10.4 to 1.9]

2. Secondary Outcome: Expert Panel Scar Assessment Score at Week 24: Part B
Description: Scar assessment by an expert panel was done on blinded photographs using 100 mm VAS where a score of 0 = best possible scar and a score of 100 = worst possible scar. A pair of photographs for each participant was presented and evaluated 3 times by an expert panel.
Time Frame: Week 24
Population: Completer population included all participants who had missed not more than 1 dose of study drug, had the Week 12 assessment and non-missing data for VAS scar assessment score. Here 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeter
Arm/Group | EXC 001 (PF-0647387) During Part B | Placebo During Part B
Number analyzed (Participants) | 31 | 31
millimeter | 37.9 (9.29) | 37.6 (10.73)
Statistical Analysis 1: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.858, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-3.5 to 4.2]

3. Secondary Outcome: Physician Observer Scar Assessment Score at Week 12 and 24: Part B
Description: Physician assessment of scar was done using a valid published 10-point rating scale. Physician rated vascularity, pigmentation, thickness, relief, pliability, surface area and overall opinion for a scar on a score of 1 = normal skin to 10 = worst scar imaginable. Composite score was the sum of all the scores except the overall opinion score and range from 6 (best score) to 60 (worst score).
Time Frame: Week 12 and 24
Population: Completer population included all participants who had missed not more than 1 dose of study drug, had the Week 12 assessment and non-missing data for VAS scar assessment score. Here 'n' signifies those participants who were evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 (PF-0647387) During Part B | Placebo During Part B
Number analyzed (Participants) | 32 | 32
units on a scale
  Week 12: Vascularity | 3.7 (1.49) | 4.7 (1.69)
  Week 12: Pigmentation | 3.2 (1.40) | 3.7 (1.63)
  Week 12: Thickness | 3.2 (1.52) | 4.6 (1.95)
  Week 12: Relief | 2.8 (1.36) | 3.7 (1.84)
  Week 12: Pliability | 2.9 (1.50) | 3.7 (1.68)
  Week 12: Surface Area | 3.7 (1.77) | 4.1 (1.62)
  Week 12: Overall Opinion | 3.5 (1.59) | 4.4 (1.56)
  Week 12: Composite Score | 19.5 (7.10) | 24.5 (8.10)
  Week 24: Vascularity: number analyzed (Participants) | 31 | 31
  Week 24: Vascularity | 3.3 (1.27) | 3.2 (1.34)
  Week 24: Pigmentation: number analyzed (Participants) | 31 | 31
  Week 24: Pigmentation | 3.6 (1.58) | 3.2 (1.45)
  Week 24: Thickness: number analyzed (Participants) | 31 | 31
  Week 24: Thickness | 3.3 (1.47) | 3.5 (1.48)
  Week 24: Relief: number analyzed (Participants) | 31 | 31
  Week 24: Relief | 2.6 (1.48) | 2.6 (1.43)
  Week 24: Pliability: number analyzed (Participants) | 31 | 31
  Week 24: Pliability | 2.7 (1.67) | 2.7 (1.60)
  Week 24: Surface Area: number analyzed (Participants) | 31 | 31
  Week 24: Surface Area | 3.4 (1.50) | 3.4 (1.56)
  Week 24: Overall Opinion: number analyzed (Participants) | 31 | 31
  Week 24: Overall Opinion | 3.3 (1.16) | 3.3 (1.37)
  Week 24: Composite Score: number analyzed (Participants) | 31 | 31
  Week 24: Composite Score | 19.0 (8.01) | 18.5 (7.88)
Statistical Analysis 1: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Vascularity: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -1.0, 95% CI 2-sided [-1.6 to -0.4]
Statistical Analysis 2: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Pigmentation: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.067, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.1 to 0.0]
Statistical Analysis 3: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Thickness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-2.1 to -0.7]
Statistical Analysis 4: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Relief: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.002, t-test, 2 sided; Median Difference (Final Values) = -0.9, 95% CI 2-sided [-1.4 to -0.4]
Statistical Analysis 5: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Pliability: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.007, t-test, 2 sided; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.3 to -0.2]
Statistical Analysis 6: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Surface Area: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.214, t-test, 2 sided; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.1 to 0.3]
Statistical Analysis 7: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Overall Opinion: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.003, t-test, 2 sided; Mean Difference (Final Values) = -0.9, 95% CI 2-sided [-1.5 to -0.3]
Statistical Analysis 8: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = -5.0, 95% CI 2-sided [-7.8 to -2.2]
Statistical Analysis 9: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Vascularity: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.673, t-test, 2 sided; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.5 to 0.7]
Statistical Analysis 10: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Pigmentation: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.276, t-test, 2 sided; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.3 to 1.1]
Statistical Analysis 11: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Thickness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.670, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.5]
Statistical Analysis 12: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Relief: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 1.000, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.5]
Statistical Analysis 13: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Pliability: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.909, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 14: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Surface Area: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.852, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.6 to 0.8]
Statistical Analysis 15: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Overall Opinion: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.906, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.5 to 0.6]
Statistical Analysis 16: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.768, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-2.8 to 3.8]

4. Secondary Outcome: Participants Observer Scar Assessment Score at Week 12 and 24: Part B
Description: Participants rated pain, itching, color, stiffness, thickness, irregularity, and overall opinion of scar on 10-point scale. For pain and itching associated with scar: range = 1 (no, not at all) to 10 (yes, worst imaginable) and for other parameters associated with scar compared to normal skin: range = 1 (no, same as normal skin) to 10 (yes, very different). Composite score = sum of all scores except overall opinion, range 6 (best) to 60 (worst). Scar appearance composite score = sum of all scores except overall opinion, pain and itching, range 4 (best) to 40 (worst).
Time Frame: Week 12 and 24
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | EXC 001 (PF-0647387) During Part B | Placebo During Part B
Number analyzed (Participants) | 32 | 32
units on a scale
  Week 12: Pain | 2.0 (1.50) | 1.9 (1.68)
  Week 12: Itching | 1.8 (1.35) | 1.8 (1.32)
  Week 12: Color | 5.8 (2.42) | 6.5 (2.49)
  Week 12: Stiffness | 4.3 (2.21) | 4.4 (2.00)
  Week 12: Thickness | 4.3 (2.37) | 4.7 (2.54)
  Week 12: Irregular | 4.7 (2.46) | 5.3 (2.44)
  Week 12: Overall Opinion | 4.3 (1.97) | 5.0 (2.18)
  Week 12: Composite Score | 22.9 (7.34) | 24.7 (7.44)
  Week 12: Scar Appearance Composite Score | 19.1 (6.87) | 20.9 (7.27)
  Week 24: Pain: number analyzed (Participants) | 31 | 31
  Week 24: Pain | 1.4 (1.05) | 1.1 (0.34)
  Week 24: Itching: number analyzed (Participants) | 31 | 31
  Week 24: Itching | 1.7 (1.60) | 1.5 (1.46)
  Week 24: Color: number analyzed (Participants) | 31 | 31
  Week 24: Color | 6.3 (2.44) | 5.8 (2.70)
  Week 24: Stiffness: number analyzed (Participants) | 31 | 31
  Week 24: Stiffness | 3.8 (1.80) | 4.3 (2.52)
  Week 24: Thickness: number analyzed (Participants) | 31 | 31
  Week 24: Thickness | 4.1 (2.33) | 4.1 (2.35)
  Week 24: Irregular: number analyzed (Participants) | 31 | 31
  Week 24: Irregular | 4.9 (2.57) | 4.9 (2.78)
  Week 24: Overall Opinion: number analyzed (Participants) | 31 | 31
  Week 24: Overall Opinion | 4.7 (2.14) | 4.8 (2.50)
  Week 24: Composite Score: number analyzed (Participants) | 31 | 31
  Week 24: Composite Score | 22.1 (8.61) | 21.8 (9.65)
  Week 24: Scar Appearance Composite Score: number analyzed (Participants) | 31 | 31
  Week 24: Scar Appearance Composite Score | 19.1 (8.06) | 19.2 (8.97)
Statistical Analysis 1: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12 Pain: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.773, t-test, 2 sided; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.4 to 0.5]
Statistical Analysis 2: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Itching: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 1.000, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.4 to 0.4]
Statistical Analysis 3: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Color: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.072, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.4 to 0.1]
Statistical Analysis 4: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Stiffness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.851, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.6]
Statistical Analysis 5: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Thickness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.184, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.2 to 0.2]
Statistical Analysis 6: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Irregular: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.059, t-test, 2 sided; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-1.3 to 0.0]
Statistical Analysis 7: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Overall Opinion: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.040, t-test, 2 sided; Mean Difference (Final Values) = -0.8, 95% CI 2-sided [-1.5 to -0.0]
Statistical Analysis 8: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.120, t-test, 2 sided; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-4.1 to 0.5]
Statistical Analysis 9: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 12, Scar Appearance Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.094, t-test, 2 sided; Mean Difference (Final Values) = -1.8, 95% CI 2-sided [-4.0 to 0.3]
Statistical Analysis 10: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Pain: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.243, t-test, 1 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 11: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Itching: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.339, t-test, 2 sided; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6]
Statistical Analysis 12: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Color: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.250, t-test, 2 sided; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.3 to 1.2]
Statistical Analysis 13: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Stiffness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.164, t-test, 2 sided; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.3 to 0.2]
Statistical Analysis 14: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Thickness: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 1.000, t-test, 2 sided; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.8 to 0.8]
Statistical Analysis 15: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Irregular: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.928, t-test, 2 sided; Mean Difference (Final Values) = -0.0, 95% CI 2-sided [-0.8 to 0.7]
Statistical Analysis 16: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Overall Opinion: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.865, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.8 to 0.7]
Statistical Analysis 17: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.804, t-test, 2 sided; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-2.3 to 3.0]
Statistical Analysis 18: Comparison: EXC 001 (PF-0647387) During Part B vs Placebo During Part B; Week 24, Scar Appearance Composite Score: Comparison within the participant between EXC 001 and placebo; Test type: Superiority; p = 0.937, t-test, 2 sided; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.6 to 2.4]

5. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. AEs included SAEs and all non-SAEs that occurred during the study.
Time Frame: Day 1 of Part A up to Week 24 of Part B
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- EXC 001 (PF-0647387) During Part A: In Part A participants received single intradermal injections on lower back of EXC 001 at a dose of 5 mg on Day 1 and 21. Third 5 mg intradermal injection of EXC 001 was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery (Day 1 in Part B). The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until day of surgery in Part B.
- EXC 001 (PF-0647387) + Placebo During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent abdominoplasty surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of abdominoplasty incision on one side of the midline and 4 intradermal injections of placebo matched to EXC 001 to a 6 cm section of both sides of abdominoplasty incision on another side of the midline, at Week 2, 5, 8, and 11 after the surgical incision was closed.
Arm/Group | EXC 001 (PF-0647387) During Part A | EXC 001 (PF-0647387) + Placebo During Part B
Number analyzed (Participants) | 41 | 33
Participants
  AEs | 7 | 21
  SAEs | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormal Physical Examinations Findings: Part A and Part B
Description: Physical examination included the assessment of skin; head, ears, eyes, nose, and throat; respiratory; cardiovascular; abdomen; musculoskeletal; neurological; gastrointestinal; genitourinary; endocrine and lymph nodes. Abnormal physical examinations findings was based on investigator's discretion.
Time Frame: Day 1 of Part A up to Week 12 of Part B
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-0647387) During Part A | EXC 001 (PF-0647387) + Placebo During Part B
Number analyzed (Participants) | 41 | 33
Participants | 3 | 3

7. Secondary Outcome: Number of Participants With Clinically Significant Findings in Electrocardiogram (ECG): Part A and Part B
Description: Number of participants with clinically significant abnormality in ECG were reported. Clinical significance was based on investigator's discretion.
Time Frame: Day 1 of Part A up to Week 12 of Part B
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-0647387) During Part A | EXC 001 (PF-0647387) + Placebo During Part B
Number analyzed (Participants) | 41 | 33
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Findings in Laboratory Examinations: Part A and Part B
Description: Laboratory analysis included hematology, biochemistry and urinalysis. Hematology range: basophils (bas) 0-0.2, eosinophils (eos) 0-0.4, leukocytes (leu) 4-10.5, lymphocytes (lym) 0.7-4.5, neutrophils (neu) 1.8-7.8, platelet 140-415, monocytes (mon) 0.1-1 in 10^9 per liter; bas/leu 0-3, eos/leu 0-7, lym/leu 14-46, mon/leu 4-13, neu/leu and neu/leu 40-74 in percentage, erythrocytes 3.8-5.1 10^12/L, hematocrit 0.34-0.44 L/L, hemoglobin 115-150 gram per liter (g/L). Biochemistry range: creatine kinase 24-173, alkaline phosphatase 25-150, alanine aminotransferase (AT) and aspartate AT 0-40 in International units per liter; creatinine 50-88, urate 89-399, bilirubin 2-21 in micromole per liter, glucose 3.6-5.5, potassium 3.5-5.5, sodium 135-148, blood urea nitrogen 1.8-9.3 in millimole/L, albumin 35-55 g/L. Urinalysis parameters: pH (5-7.5), specific gravity (1.005-1.03). Participants with clinically significant findings were reported.
Time Frame: Day 1 of Part A up to Week 12 of Part B
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- EXC 001 (PF-0647387) During Part A: In Part A participants received 2 intradermal injections on lower back of EXC 001 at a dose of 5 mg on Day 1 and 21. Third 5 mg intradermal injection of EXC 001 was administered at the discretion of Investigator based on the event of an equivocal skin sensitization on Day 38 or at least 7 days prior to surgery (Day 1 in Part B). The injection site was evaluated immediately after the injection and on Days 21, 28, 38, 50 until day of surgery in Part B.
Arm/Group | EXC 001 (PF-0647387) During Part A | EXC 001 (PF-0647387) + Placebo During Part B
Number analyzed (Participants) | 41 | 33
Participants | 0 | 2

9. Secondary Outcome: Number of Participants With Clinically Significant Findings in Vital Signs and Weight: Part A and Part B
Description: Following vital sign parameters were assessed: diastolic blood pressure, systolic blood pressure, respiration rate, pulse rate, and temperature. Number of participants with clinically significant change in any vital sign parameter and weight compared to baseline were reported. Clinical significance was based on investigator's discretion.
Time Frame: Day 1 of Part A up to Week 12 of Part B
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-0647387) During Part A | EXC 001 (PF-0647387) + Placebo During Part B
Number analyzed (Participants) | 41 | 33
Participants | 0 | 0

10. Secondary Outcome: Number of Participants With Positive Skin Sensitivity Reaction: Part A and Part B
Description: Participants were instructed to inform the investigator in case of any itching, redness, pain or any other symptom that appears to be a rash at the injection sites. Erythematous, raised (indurated) and edematous reactions were considered as positive skin sensitivity reactions.
Time Frame: Day 21 of Part A up to Day 14 of Part B
Population: Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | EXC 001 (PF-0647387) During Part A | EXC 001 (PF-0647387) + Placebo During Part B
Number analyzed (Participants) | 41 | 33
Participants | 0 | 4

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Safety population included participants who completed Day 1 of Part A and received at least 1 dose of study drug. Safety assessment was not planned separately for EXC 001 and placebo.
Groups:
- Active Dosing Phase During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants underwent abdominoplasty surgery on Day 1 and then received 4 intradermal injections of EXC 001 at dose of 5 mg per linear cm to a 6 cm section of both sides of abdominoplasty incision on one side of the midline at Week 2, 5, 8, and 11 after the surgical incision was closed. Active dosing phase was from Week 2 to Week 13.
- Post Dosing Phase During Part B: Participants who tested negative for skin sensitization in Part A were eligible for Part B. In Part B, participants who received treatment in active dosing phase were followed up from Week 13 until end of the study in post dosing phase.
Arm/Group | EXC 001 (PF-0647387) During Part A | Active Dosing Phase During Part B | Post Dosing Phase During Part B
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/33 | 0/32
Other Adverse Events (participants affected / at risk) | 7/41 | 18/33 | 3/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | EXC 001 (PF-0647387) During Part A (N=41) | Active Dosing Phase During Part B (N=33) | Post Dosing Phase During Part B (N=32)
Nasopharyngitis (Infections and infestations) | 1 | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 0 | 1 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0
Vaginitis bacterial (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract (Infections and infestations) | 0 | 1 | 0
Incision site pruritus (Injury, poisoning and procedural complications) | 0 | 3 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 0
Suture rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0
Injection site erythema (General disorders) | 0 | 2 | 0
Cyst (General disorders) | 0 | 1 | 0
Infusion site rash (General disorders) | 0 | 1 | 0
Injection site pruritus (General disorders) | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.